CLINICAL TRIAL: NCT00000134
Title: Cytomegalovirus Retinitis Retreatment Trial
Brief Title: Studies of the Ocular Complications of AIDS (SOCA)--Cytomegalovirus Retinitis Retreatment Trial (CRRT)
Acronym: CRRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Eye Institute (NEI) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Johns Hopkins University (Other); University of Wisconsin, Madison (Other); Baylor College of Medicine (Other); Tulane University School of Medicine (Other); Icahn School of Medicine at Mount Sinai (Other); New York Presbyterian Hospital (Other); New York University (Other); Northwestern University (Other); University of California, Los Angeles (Other); University of California, San Francisco (Other); University of California, San Diego (Other); University of Miami (Other); University of North Carolina, Chapel Hill (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Curtis Meinert, Curtis Meinert, PhD, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-33; U10EY008057 (NIH); U01AI027668 (NIH)
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Results first posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-08

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome; Cytomegalovirus Retinitis
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Cytomegalovirus Retinitis | interventions — Ganciclovir; Foscarnet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- intravenous foscarnet (Experimental): intravenous foscarnet reinduction at 90 mg/kg twice daily for 2 weeks, followed by maintenance therapy at 120 mg/kg/day
  Interventions: Drug: Foscarnet
- intravenous ganciclovir (Active Comparator): intravenous ganciclovir reinduction at 5 mg/kg twice daily for 2 weeks followed by maintenance at 10 mg/kg/day
  Interventions: Drug: Ganciclovir
- combination therapy (Active Comparator): combination therapy, wherein patients continued their previous therapy and were reinduced with the second drug and then placed on maintenance therapy with foscarnet at 90 mg/kg/day and ganciclovir at 5 mg/kg/day.
  Interventions: Drug: Ganciclovir; Drug: Foscarnet

INTERVENTIONS:
Drug: Ganciclovir — intravenous ganciclovir induction at 5 mg/kg twice daily for 2 weeks followed by maintenance at 10 mg/kg/day
  Other Names: cytovene
  Arms: combination therapy; intravenous ganciclovir
Drug: Foscarnet — intravenous foscarnet induction at 90 mg/kg twice daily for 2 weeks, followed by maintenance therapy at 120 mg/kg/day
  Other Names: foscavir
  Arms: combination therapy; intravenous foscarnet

SUMMARY:
To compare the relative merits of three therapeutic regimens in patients with AIDS and CMV retinitis who have been previously treated but whose retinitis either is nonresponsive or has relapsed. These three therapeutic regimens were (1) foscarnet, (2) high-dose ganciclovir, and (3) combination foscarnet and ganciclovir.

To compare two treatment strategies in patients with relapsed or nonresponsive CMV retinitis: (1) continuing the same anti-CMV drug or (2) switching to the alternate drug.

DETAILED DESCRIPTION:
CMV retinitis is the most common intraocular infection in patients with AIDS and is estimated to affect 35 to 40 percent of patients with AIDS. Untreated CMV retinitis is a progressive disorder, the end result of which is total retinal destruction and blindness. At the time of this trial, drugs approved by the United States Food and Drug Administration (FDA) for the treatment of CMV retinitis were ganciclovir (Cytovene) and foscarnet (Foscavir). Although most retinitis responds well to initial therapy with systemically administered drugs, given enough time, nearly all patients will suffer a relapse of the retinitis. Relapsed retinitis generally responds to reinduction and maintenance therapy, but the interval between successive relapses progressively shortens. The CRRT addressed the issue of the management of relapsed CMV retinitis.

The CRRT was a multicenter, randomized, controlled clinical trial comparing three regimens in patients with relapsed retinitis. Patients with AIDS and CMV retinitis that had relapsed or was nonresponsive to initial therapy were randomized to one of three regimens: (1) intravenous foscarnet reinduction at 90 mg/kg twice daily for 2 weeks, followed by maintenance therapy at 120 mg/kg/day; (2) intravenous ganciclovir reinduction at 5 mg/kg twice daily for 2 weeks followed by maintenance at 10 mg/kg/day; and (3) combination therapy, wherein patients continued their previous therapy and were reinduced with the second drug and then placed on maintenance therapy with foscarnet at 90 mg/kg/day and ganciclovir at 5 mg/kg/day.

ELIGIBILITY:
inclusion criteria: Males and females eligible for the CRRT must have been age 18 years or older and have had AIDS and CMV retinitis. They must have had active CMV despite a minimum of 28 days of previous treatment with an anti-CMV drug. Furthermore, they must have had an absolute neutrophil count greater than or equal to 500 cells/µL, platelet count greater than or equal to 20,000 cells/µL, and a serum creatinine < 2.5 mg/dL in order to tolerate the drug regimens.

exclusion criteria: history of intolerance to ganciclovir or foscarnet, history of therapy involving the combination of foscarnet and ganciclovir, unwillingness to practice appropriate birth control, active drug or alcohol abuse, media opacity, retinal detachment not scheduled for surgical repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 1992-12; Primary Completion 1995-03 (Actual); Study Completion 1995-03 (Actual)

REFERENCES:
- [Background] Combination foscarnet and ganciclovir therapy vs monotherapy for the treatment of relapsed cytomegalovirus retinitis in patients with AIDS. The Cytomegalovirus Retreatment Trial. The Studies of Ocular Complications of AIDS Research Group in Collaboration with the AIDS Clinical Trials Group. Arch Ophthalmol. 1996 Jan;114(1):23-33. doi: 10.1001/archopht.1996.01100130021004. PMID 8540847
- [Background] Martin BK, Kaplan Gilpin AM, Jabs DA, Wu AW; Studies of Ocular Complications of AIDS Research Group. Reliability, validity, and responsiveness of general and disease-specific quality of life measures in a clinical trial for cytomegalovirus retinitis. J Clin Epidemiol. 2001 Apr;54(4):376-86. doi: 10.1016/s0895-4356(00)00294-8. PMID 11305288

RESULTS

PARTICIPANT FLOW:
Recruitment Details: December 1992
Period: Overall Study
Arm/Group | Intravenous Foscarnet | Intravenous Ganciclovir | Combination Therapy
Started | 89 | 94 | 96
Completed | 89 | 94 | 96
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Foscarnet | Intravenous Ganciclovir | Combination Therapy | Total
Number analyzed (Participants) | 89 | 94 | 96 | 279
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 89 | 94 | 96 | 279
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 10 | 23
  Male | 82 | 88 | 86 | 256
Region of Enrollment [Number; unit: participants]
  United States | 89 | 94 | 96 | 279

OUTCOME MEASURES:

1. Primary Outcome: Morbidity
Description: To determine the best therapeutic regimen, using currently approved drugs, for treatment of relapsed cytomegalovirus (CMV) retinitis.
Time Frame: Patients will be seen at baseline, monthly for six months, and then every three months until death or termination of the trial
Measure: Number; unit: participants
Arm/Group | Intravenous Foscarnet | Intravenous Ganciclovir | Combination Therapy
Number analyzed (Participants) | 88 | 93 | 93
participants | 88 | 93 | 93

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Arm/Group | Intravenous Foscarnet | Intravenous Ganciclovir | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 32/88 | 41/93 | 51/93
Other Adverse Events (participants affected / at risk) | 7/88 | 7/93 | 10/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Foscarnet (N=88) | Intravenous Ganciclovir (N=93) | Combination Therapy (N=93)
Neutropenia (Blood and lymphatic system disorders) | 32 (86) | 41 (95) | 51 (107)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (28) | 8 (19) | 15 (40)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Foscarnet (N=88) | Intravenous Ganciclovir (N=93) | Combination Therapy (N=93)
Hospitalizations (Infections and infestations) | 7 (9) | 7 (10) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days